CLINICAL TRIAL: NCT05540054
Title: Investigation of Inspiratory Muscle Training Efficiency Before Bronchoscopic Procedure in Chronic Obstructive Pulmonary Diseases
Brief Title: Inspiratory Muscle Training Efficiency Before Bronchoscopic Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLVR_IMT
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2022-09

CONDITIONS: Copd; IMT
Keywords: IMT; COPD; pulmonary rehabilitation; bronchoscopic procedure; Bronchoscopic lung volume reduction; valve; coil; balloon
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pulmonary rehabilitation group (PR) (Experimental): Patients diagnosed with COPD and listed for bronchoscopic procedure.
  Interventions: Other: Standard pulmonary rehabilitation programme
- Inspiratory muscle training group (PR+IMT) (Experimental): Patients diagnosed with COPD and listed for bronchoscopic procedure.
  Interventions: Other: Inspiratory muscle training; Other: Standard pulmonary rehabilitation programme

INTERVENTIONS:
Other: Inspiratory muscle training — Respiratory muscle strengthening training will be given with a resistive threshold inspiratory muscle strengthening device.
  Arms: Inspiratory muscle training group (PR+IMT)
Other: Standard pulmonary rehabilitation programme — The standard PR consisted of breathing exercises, peripheral muscle strengthening and self walking training.

SUMMARY:
The aim of this study is to examine the effectiveness of inspiratory muscle training (IMT) before bronchoscopic procedure in Chronic Obstructive Pulmonary Patients (COPD). Patients with a diagnosis of COPD, who are listed for a bronchoscopic procedure and referred to the pulmonary rehabilitation (PR) clinic, will be randomly divided into two groups. Standard PR exercise program will be applied to both groups. In addition to the standard program, IMT will be applied to one of the groups. The effect of IMT on exercise program gains will be examined.

DETAILED DESCRIPTION:
* Cases diagnosed with COPD by a chest diseases specialist at Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital will be included in the study.
* The cases meeting the inclusion criteria will be randomized and divided into two groups, called the standard rehabilitation group (PRGr) and the inspiratory muscle training group (IMTGr).
* Initial exercise sessions and all evaluations of all cases will be performed in the hospital. The 2nd and 3rd training repetitions will be held at their homes via online synchronized videoconferencing. The exercise video will be sent to the smart phones of the cases who have completed 3 training sessions. Participants will be called once a week by phone and exercise follow-up will be carried out.
* All subjects will continue to exercise 5 days a week for 2 months. The standard PR consists of breathing exercises, peripheral muscle strength and self walking training. In addition, IMT was applied to IMTGr.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-75
* Having a diagnosis of COPD diagnosed according to clinical diagnostic criteria according to -American Thoracic and European Respiratory Societies (ATS-ERS) and being a candidate patient for bronchoscopic lung volume reduction procedure
* Presence of dyspnea on exertion
* Stable clinical state at the time of inclusion without infection or exacerbation in the previous 4 weeks
* Ability to use a smart phone

Exclusion Criteria:

* Patients with severe comorbid diseases, unstable coronary artery disease, collagen vascular diseases and needing high flow oxygen therapy (˃ 3-4 L \min).
* A history of effort-related syncope or any comorbidity (such as severe orthopedic or neurological deficits or unstable heart disease) that precludes exercise training.
* Participation in a pulmonary rehabilitation program within the past 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | Change from baseline at 2 months
  The 6-minute walking test will conduct in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines. Participants will ask to walk as far as they can. Prior to and following the test, oxygen saturation, heart rate and Borg fatigue rating will measure, and the walking distance will record.
Dyspnea perception | Change from baseline at 2 months
  Modified Medical Council Dyspnea score will rate the sensation of dyspnea as the person perceives it.The severity of dyspnea is rated on a scale of 0 to 4."0 point" means no dyspnea perception and "4point" means severe dyspnea perception.
Respiratory muscle strength | Change from baseline at 2 months
  The mouth pressure measurement (maximum inspiratory and expiratory pressure) will perform with the Pony Fx spirometry device. Patient will place a rubber mouthpiece with flanges, on the device, exhale/inhale slowly and completely, and then will try to breath in as hard as possible. The patient will allow to rest for about a minute and the maneuver will repeat. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value will obtain.
Clinical status follow-up after bronchoscopic procedure | Change from baseline at 1 year after bronchoscopic procedure
  Complications and clinical status will be followed up for 1 year after the bronchoscopic procedure.

SECONDARY OUTCOMES:
Fatigue severity | Change from baseline at 2 months
  The fatigue severity scale: A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity.
Physical activity level | Change from baseline at 2 months
  The International Physical Activity Questionnaire (IPAQ) was developed as an instrument for cross-national monitoring of physical activity and inactivity. This measure assesses the types of intensity of physical activity and sitting time that people do as part of daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.
Anxiety level | Change from baseline at 2 months
  Hospital Anxiety Depression scale:The levels of anxiety will asses by Hospital Anxiety Depression Scale (HADS) .The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).Several studies suggest a cut-off score of ≥8 to be optimal for best sensitivity and specificity. The HADS has sensitivity and specificity of about 80%, and a predictive validity for identification of about 70%.
Depression level | Change from baseline at 2 months
  Hospital Anxiety Depression scale:The levels of depression will asses by Hospital Anxiety Depression Scale (HADS) .The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).Several studies suggest a cut-off score of ≥8 to be optimal for best sensitivity and specificity. The HADS has sensitivity and specificity of about 80%, and a predictive validity for identification of about 70%.
Quality of life level | Change from baseline at 2 months
  Saint George Respiratory Questionaire (SGRQ) score: The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
Pulmonary function tests (PFTs) | Change from baseline at 2 months
  PFTs will perform by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines
Peripheral muscle strength measurement | Change from baseline at 2 months
  Peripheral muscle strength measurement will be performed on major muscle groups (quadriceps femoris, tibialis anterior, iliopsoas, biceps brachii, triceps, hand grip force) with a digital muscle strength measurement device.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehlivan, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided